CLINICAL TRIAL: NCT05504681
Title: Integration of Neurocognitive Biomarkers Into a Neuro-Oncology Clinic
Status: Recruiting | Type: Observational
Sponsor: Baptist Health South Florida (Other)
Collaborators: Brainlab AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-KOT-004
Record Dates: First submitted 2022-04-08; First posted 2022-08-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Neurocognitive Disorders
Keywords: Neurocognitive; Brainlab Cognition app
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — It takes the patient on average 15 minutes to complete the Brainlab Cognition app.

SUMMARY:
This is prospective observational registry study that will assess 1) if the neurocognitive function app (Brainlab Cognition) can be used in a widespread neuro-oncology clinic setting and 2) if patient reported quality of life parameters can be obtained electronically and integrated into clinic.

ELIGIBILITY:
Inclusion Criteria:

1. All adult (18+) patients with central nervous system (CNS) tumors, both primary brain malignancies and brain metastases, treated with radiotherapy (partial brain, stereotactic radiosurgery, stereotactic fractionated radiotherapy, or whole-brain radiotherapy), surgery, and/or antineoplastic therapy and followed thereafter at Miami Cancer Institute (MCI)
2. Life expectancy ≥ 6 months
3. Willingness to participate in ongoing registration study

Exclusion Criteria:

1. Patients receiving radiotherapy to the brain for functional disease (arteriovenous malformations, trigeminal neuralgia, essential tremors, etc.)
2. Pediatric patients (<18 years old), pregnant women, and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (18+) patients with CNS tumors, both primary brain malignancies and brain metastases, treated with radiotherapy (partial brain, stereotactic radiosurgery, stereotactic fractionated radiotherapy, or whole-brain radiotherapy), surgery, and/or antineoplastic therapy and followed thereafter at Miami Cancer Institute (MCI).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Learning and memory (Neurocognitive Decline) | Baseline, 2, 4, 6, 12, 18, 24 months
  Learning and memory will be assessed by the number of correct responses (the total number of words correctly recalled). The "Verbal Recall" test will be used to measure the number of correct responses over 3 trials, the "Verbal Revision" will be used to measure the number of total correct responses, and the "Verbal Recognition" test will be used to measure number of correct responses minus the incorrect responses. Change is calculated as baseline score subtracted from post-baseline score over time.
Change in Attention and Speed of Processing (Neurocognitive Decline) | Baseline, 2, 4, 6, 12, 18, 24 months
  This will be measured by the "Symbols Matching" test. Subjects will be asked to match symbols and corresponding numbers during 90 seconds. The score will be calculated by totaling the number of correct answers during the allotted time. A higher score indicates better functioning.
Change in Verbal Fluency (Neurocognitive Decline) | Baseline, 2, 4, 6, 12, 18, 24 months
  This will be measured by the "Words That Start With" test. The total number of words correctly generated (no numbers, no proper names) by the subject will be recorded to generate their score. A higher score indicates better functioning.
Change in Fine motor and speed (Neurocognitive Decline) | Baseline, 2, 4, 6, 12, 18, 24 months
  This will be measured by the "Numbers Ordering" test. This test assesses visual scanning and motor tracking requiring focused attention. Subjects are required to sequentially connect numbered dots in ascending order that are randomly scattered on the screen in consecutive order. The total time in seconds to complete the array will be recorded as the score result. A lower score indicates better functioning.
Change in Executive functions (Neurocognitive Decline). | Baseline, 2, 4, 6, 12, 18, 24 months
  This will be measured by "Numbers and Letters Ordering" test. This test includes a divided attention component requiring mental flexibility (i.e., executive function). On this subtest, dots with numbers and letters are randomly scattered. Subjects are required to alternate between connecting numbers and letters in an ascending sequential order. Subjects will order numbers and letters from 1 to 13 and from A to M by tapping them as fast as possible in consecutive and alternating order. The total time in whole seconds to complete the array will be recorded. A lower score indicates better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh R Kotecha, MD, Principal Investigator — Miami Cancer Institute
Locations (1):
- Miami Cancer Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wefel JS, Vardy J, Ahles T, Schagen SB. International Cognition and Cancer Task Force recommendations to harmonise studies of cognitive function in patients with cancer. Lancet Oncol. 2011 Jul;12(7):703-8. doi: 10.1016/S1470-2045(10)70294-1. Epub 2011 Feb 25. PMID 21354373
- [Background] Noll KR, Bradshaw ME, Rexer J, Wefel JS. Neuropsychological Practice in the Oncology Setting. Arch Clin Neuropsychol. 2018 May 1;33(3):344-353. doi: 10.1093/arclin/acx131. PMID 29718081
- [Background] Horowitz TS, Suls J, Trevino M. A Call for a Neuroscience Approach to Cancer-Related Cognitive Impairment. Trends Neurosci. 2018 Aug;41(8):493-496. doi: 10.1016/j.tins.2018.05.001. Epub 2018 Jun 12. PMID 29907436
- [Background] Armstrong TS, Wefel JS, Wang M, Gilbert MR, Won M, Bottomley A, Mendoza TR, Coens C, Werner-Wasik M, Brachman DG, Choucair AK, Mehta M. Net clinical benefit analysis of radiation therapy oncology group 0525: a phase III trial comparing conventional adjuvant temozolomide with dose-intensive temozolomide in patients with newly diagnosed glioblastoma. J Clin Oncol. 2013 Nov 10;31(32):4076-84. doi: 10.1200/JCO.2013.49.6067. Epub 2013 Oct 7. PMID 24101048
- [Background] Gilbert MR, Dignam JJ, Armstrong TS, Wefel JS, Blumenthal DT, Vogelbaum MA, Colman H, Chakravarti A, Pugh S, Won M, Jeraj R, Brown PD, Jaeckle KA, Schiff D, Stieber VW, Brachman DG, Werner-Wasik M, Tremont-Lukats IW, Sulman EP, Aldape KD, Curran WJ Jr, Mehta MP. A randomized trial of bevacizumab for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):699-708. doi: 10.1056/NEJMoa1308573. PMID 24552317
- [Background] Lange M, Joly F, Vardy J, Ahles T, Dubois M, Tron L, Winocur G, De Ruiter MB, Castel H. Cancer-related cognitive impairment: an update on state of the art, detection, and management strategies in cancer survivors. Ann Oncol. 2019 Dec 1;30(12):1925-1940. doi: 10.1093/annonc/mdz410. PMID 31617564
- [Background] Brown PD, Pugh S, Laack NN, Wefel JS, Khuntia D, Meyers C, Choucair A, Fox S, Suh JH, Roberge D, Kavadi V, Bentzen SM, Mehta MP, Watkins-Bruner D; Radiation Therapy Oncology Group (RTOG). Memantine for the prevention of cognitive dysfunction in patients receiving whole-brain radiotherapy: a randomized, double-blind, placebo-controlled trial. Neuro Oncol. 2013 Oct;15(10):1429-37. doi: 10.1093/neuonc/not114. Epub 2013 Aug 16. PMID 23956241
- [Background] Gondi V, Pugh SL, Tome WA, Caine C, Corn B, Kanner A, Rowley H, Kundapur V, DeNittis A, Greenspoon JN, Konski AA, Bauman GS, Shah S, Shi W, Wendland M, Kachnic L, Mehta MP. Preservation of memory with conformal avoidance of the hippocampal neural stem-cell compartment during whole-brain radiotherapy for brain metastases (RTOG 0933): a phase II multi-institutional trial. J Clin Oncol. 2014 Dec 1;32(34):3810-6. doi: 10.1200/JCO.2014.57.2909. Epub 2014 Oct 27. PMID 25349290
- [Background] Casey DL, Pitter KL, Kushner BH, Cheung NV, Modak S, LaQuaglia MP, Wolden SL. Radiation Therapy to Sites of Metastatic Disease as Part of Consolidation in High-Risk Neuroblastoma: Can Long-term Control Be Achieved? Int J Radiat Oncol Biol Phys. 2018 Apr 1;100(5):1204-1209. doi: 10.1016/j.ijrobp.2018.01.008. Epub 2018 Jan 9. PMID 29439882
- [Background] De Ruysscher D, Niedermann G, Burnet NG, Siva S, Lee AWM, Hegi-Johnson F. Radiotherapy toxicity. Nat Rev Dis Primers. 2019 Feb 21;5(1):13. doi: 10.1038/s41572-019-0064-5. PMID 30792503